CLINICAL TRIAL: NCT00975377
Title: Clipping vs. No Hair Removal and the Risk of Surgical Site Infection: A Randomized, Assessor Blinded Non-inferiority Clinical Trial Among Patients Undergoing General Surgical Procedures at a Community Hospital
Brief Title: Clipping Versus No Hair Removal and the Risk of Surgical Site Infections
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gundersen Lutheran Medical Foundation (Other)
Collaborators: Gundersen Lutheran Health System (Other)
Responsible Party: Principal Investigator, Kara Kallies, Advanced Research Associate under direction of Todd Kowalski, MD (PI), Gundersen Lutheran Medical Foundation
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2-09-05-001
Record Dates: First submitted 2009-09-10; First posted 2009-09-11 (Estimated); Last update posted 2015-09-07 (Estimated); Status verified 2015-09

CONDITIONS: Surgical Site Infection; Superficial Surgical Site Infection; Deep Surgical Site Infection; Organ/Space Surgical Site Infection
Keywords: hair removal; hair clipping; surgical site infection; incisional infection; wound infection
MeSH Terms: conditions — Surgical Wound Infection; Wound Infection

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- No hair removal (No Intervention): Patients randomized to the no hair removal cohort will not undergo any preoperative hair removal.
- Hair clipping (Active Comparator): Patients in the clipping cohort undergo hair removal at the surgical site. Hair removal will occur on the day of surgery immediately prior to the scheduled operation.
  Interventions: Procedure: Hair clipping

INTERVENTIONS:
Procedure: Hair clipping — Patients randomized to the hair clipping cohort will be clipped using an Allegiance 4413 hair clipper. Hair removal will occur on the day of surgery by one of the preoperative nursing staff, immediately prior to the scheduled operation.
  Arms: Hair clipping

SUMMARY:
The objective of this study is to determine whether hair clipping is non-inferior to no hair removal in preventing superficial, deep, and organ space surgical site infections (SSI) in patients undergoing various general surgical procedures, evaluated after surgery by an assessor blinded to treatment allocation. Additional goals include evaluating wound complications that arise in patients that have hair clipped and in patients that do not have hair removed and determining the impact of clipping versus no hair removal and SSI versus no SSI on length of hospital stay.

DETAILED DESCRIPTION:
Public health organizations, third party payers, consumer watchdog groups, health care quality organizations, and patients are increasingly scrutinizing patient safety in hospitals. Surgical site infection (SSI) rates are one of the key quality measures by which hospitals are evaluated. Centers for Disease Control (CDC) guidelines provide specific recommendations, weighted by evidence, to prevent SSI. These include the following category 1A recommendations (Strongly recommended for implementation and supported by well-designed experimental, clinical, or epidemiological studies).

* Do not remove hair preoperatively unless the hair at or around the incision site will interfere with the operation
* If hair is removed, remove immediately before the operation, preferably with electric clippers.

However, a recent systematic review of randomized clinical trials concluded there was no difference in SSI among patients that had hair removed prior to surgery and those that did not. Furthermore, trials involving hair removal were largely underpowered and of marginal quality. If hair is going to be removed, previous studies have shown hair removal with clippers or depilatory creams to result in fewer SSI than shaving with a razor. However, the need for trials comparing SSI rates with and without hair removal was stressed in the recent systematic review. No prospective, randomized clinical trial evaluating no hair removal vs. hair removal by clipping, the two hair removing modalities preferred by CDC SSI prevention guidelines, has ever been reported. This study aims to assess whether hair removal via clipping is non-inferior to no hair removal in a cohort of patients undergoing general surgical procedures at a community hospital.

A non-inferiority study design will be used based upon the following rationale. CDC guidelines recommend not removing hair preoperatively unless the hair will interfere with the operation. However, there is no published evidence that clipping hair results in more SSI than no hair removal. Clipping hair is often preferred from a surgical perspective. This may be because of historical practice patterns, personal comfort level, and the either real or perceived interference of unremoved hair with performing the operation. Therefore, assessing whether clipping is non-inferior to no hair removal will provide helpful information regarding the appropriateness of the current CDC recommendation to not remove hair preoperatively unless the hair will interfere with the operation.

Patients will be assessed for enrollment after a decision has been made for elective (non-emergent) operative intervention. Patients will undergo our institution's current preoperative procedural standard of care. Patients will be specifically instructed to not shave themselves prior to the procedure. The day of the procedure patients will undergo our institution's standard preoperative skin preparation, which currently includes povidone based skin antiseptic. Preoperative antibiotics will be administered according to our institutional standards of care for their particular operation.

Randomization will be assigned the day of surgery in the preoperative area. Patients will be randomized 1:1 to either undergo clipping or no hair removal. Enrolled patients will then undergo the type of hair removal appropriate for their study arm. Clipping patients will undergo hair removal on the day of surgery by a member of the preoperative nursing staff, immediately prior to the scheduled operation. Any patient that undergoes unanticipated hair removal, (either additional hair removal in patients that were clipped or any hair removal in patients that were not clipped) will be noted as a protocol deviation and the event recorded. Patients will undergo their surgical procedure according to standard surgical care.

Patients will be scheduled for a follow-up wound assessment with a trained study nurse. This assessment will take place by an independent assessor whom is blinded (as best able given study interventions) to the study group the patient was in.

Additionally, if patients are seen for wound problems by their surgeon, primary physicians, or other physicians we will attempt to have them evaluated by one of the trained nurses at that visit as well. If patients do not keep their follow-up appointment, they will be called and asked a standardized set of questions related to the wound. Finally, in the event patients are seen for wound problems at other facilities, or in other departments (i.e. urgent care, emergency room, etc), they will be encouraged to make a follow-up appointment within a few days to be reassessed, at which time the study nurse can assess their status as well. The patients' electronic medical records will be updated to reflect their study involvement, and to alert providers to contact the study coordinator with wound related questions if seen in another department.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Patients undergoing a general surgical procedure (inpatient or ambulatory)

Exclusion Criteria:

* Less than 18 years of age
* Systemic antibiotics within 1 week of surgery
* Toe amputations
* Ano-rectal surgery
* Vascular surgery
* Patients that have no need for hair to be removed for the operation
* Inability to provide consent
* Anticipated inability to keep 14 day follow-up appointment
* Emergent surgical procedure
* Patients remove their own hair prior to the operative day

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1678 (Actual)
Dates: Start 2009-10; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
To determine the proportion of patients without a surgical site infection (as defined by CDC criteria) at the postoperative assessment for patients who had hair clipped versus those with no hair removal preoperatively. | 14 (+/-7) days after surgery

SECONDARY OUTCOMES:
To evaluate the unanticipated need for antibiotic or surgical intervention of the wound, as well as wound cultures obtained and their results. | 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Todd J. Kowalski, MD, Principal Investigator — Gundersen Lutheran Health System; Shanu N. Kothari, MD, Principal Investigator — Gundersen Lutheran Health System
Locations (1):
- Gundersen Lutheran Health System, La Crosse, Wisconsin, United States

REFERENCES:
- [Background] Mangram AJ, Horan TC, Pearson ML, Silver LC, Jarvis WR. Guideline for Prevention of Surgical Site Infection, 1999. Centers for Disease Control and Prevention (CDC) Hospital Infection Control Practices Advisory Committee. Am J Infect Control. 1999 Apr;27(2):97-132; quiz 133-4; discussion 96. PMID 10196487
- [Background] Tanner J, Woodings D, Moncaster K. Preoperative hair removal to reduce surgical site infection. Cochrane Database Syst Rev. 2006 Jul 19;(3):CD004122. doi: 10.1002/14651858.CD004122.pub3. PMID 16856029
- [Derived] Kowalski TJ, Kothari SN, Mathiason MA, Borgert AJ. Impact of Hair Removal on Surgical Site Infection Rates: A Prospective Randomized Noninferiority Trial. J Am Coll Surg. 2016 Nov;223(5):704-711. doi: 10.1016/j.jamcollsurg.2016.03.032. PMID 27687471